CLINICAL TRIAL: NCT04042675
Title: The Effects of Respiratory Muscle Strength on Exercise Capacity, Fatigue and Physical Activity Level in Patients With Parkinson Disease
Brief Title: The Effects of Respiratory Muscle Strength in Parkinson Disease
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, EMEL METE, Research Assistant, Istanbul Medeniyet University
Other Study IDs: 25.07.2019/87
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; respiratuary muscle strength; physical activity level; fatigue; exercise capacity
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- parkinson group: parkinson's patients aged between 40-75 years and 1-3 according to Hoehn-Yahr stage.
  Interventions: Diagnostic Test: observational study
- Control group: healthy individuals between the ages of 40-75 and without any neurological disorders.
  Interventions: Diagnostic Test: observational study

INTERVENTIONS:
Diagnostic Test: observational study — There will be two groups in this study. One of the groups will consist of 30 parkinson's patients aged between 40-75 years and 1-3 according to Hoehn-Yahr stage. The other group will consist of 30 healthy individuals between the ages of 40-75 and without any neurological disorders. Participants' respiratory muscle strength, exercise capasity, fatigue and physical activity levels will be assessed. All asessements will done for only one time.

SUMMARY:
The aim of this study was to compare respiratory muscle strength, motor performance, fatigue and physical activity levels between patients with Parkinson disease and the healthy people and the other aim is to investigate the effects of respiratory muscle strength on exercise capasity, fatigue and physical activity levels in patients with Parkinson's disease.

There will be two groups in this study. One of the groups will consist of 30 patients aged between 40-75 years and 1-3 according to Hoehn-Yahr stage. The other group will consist of 30 healthy individuals between the ages of 40-75 and without any neurological disorders. Respiratory muscle strength, exercise capacity, fatigue and physical activity levels will be assessed.

DETAILED DESCRIPTION:
Assessment methods will include: Mouth pressure measuring for assessment of respiratory muscle strength, timed up and go (TUG) and ten meter walk test (10MWT) to assess exercise capasity, fatigue impact scale (FIS) and fatigue severity scale (FSS) to assess fatigue and the international physical activity questionnaire (IPAQ) will be used to assess physical activity levels of participants.

There will be two groups in this study. One of the groups will consist of 30 parkinson's patients aged between 40-75 years and 1-3 according to Hoehn-Yahr stage. The other group will consist of 30 healthy individuals between the ages of 40-75 and without any neurological disorders.

Including criterias:

For patients with Parkinson disease

* diagnosed with Parkinson disease
* Aged between 45-75 years
* 1-3 according to Hoehn-Yahr scale For health group
* Aged between 45-75 years
* Without any neurological disorder

Evaluation of Respiratory Muscle Strength: Maximum inspiratory (MIP) and expiratory pressures (MEP) are measurements of pressures against the closed airway to assess the strength of respiratory muscles. MIP and MEP pressures are noninvasive tests that show indirect respiratory muscle strength. Spirometry device (Carefusion /Micro RPM) will be used to assess MIP and MEP. The maximum inspiratory and expiratory valve (shutter) that closes the airway during the maximum oral pressure measured during the maximum breath.

Evaluation of Exercise Capacity: Exerise capacity of participants will assess with TUG and 10MWT tests.

Time up and go test (TUG) assesses mobility, balance, walking ability and risk of falling. The test is performed by the person getting up from a chair, walking 3 meters, turning around himself, walking back to the chair and sitting again.

Ten meter walk test (10MWT): In the test, the person is asked to walk at his / her normal speed within a pre-measured area of 10 meters. Two measurements are taken and the best value is recorded in meters per second (m / sec).

Evaluation of Fatigue: Fatigue impact scale (FIS) and Fatigue severity scale (FSS) will be used.

Fatigue impact scale (FIS) consists of forty questions. The first 10 items assess cognitive status, the second 10 items evaluate physical status, and the third 20 items evaluate psychological status. Each question is scored between 0 (no problem) and 4 (maximum problem). The highest score is 160. Higher scores show more fatigue.

Fatigue severity scale (FSS) consists of 9 questions. Each question is evaluated with a scale of 1 to 7 points. 1 = Strongly disagree, 7 = Strongly agree. Minimum score 9, maximum score 63.High scores indicate fatigue.

Evaluation of Physical Activity Level: International Physical Activiy Questionnaire (IPAQ) will be used.

The long form of the IPAQ questionnaire is used to gather information about recreational activities such as home and field activities, occupational transport, sedentary activities. The calculation of the total score for the IPAQ long form includes the sum of time (minutes) and frequency (days) for all types of activity in all areas. Scoring is done according to activity (walking, moderate activity, severe activity). From these calculations, a score in MET-minutes is obtained. A MET-minute is calculated by multiplying the minute of activity performed by the MET score. MET-min x (person's body weight kg / 60 kg).

ELIGIBILITY:
Inclusion Criteria:

For patients with Parkinson disease

* diagnosed with Parkinson disease
* Aged between 45-75 years
* 1-3 according to Hoehn-Yahr scale For health group
* Aged between 45-75 years
* Without any neurological disorder

Exclusion Criteria:

For patients with Parkinson disease

* not diagnosed with Parkinson disease
* 4-5 according to Hoehn-Yahr scale For health group
* With a neurological disorder

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons who meet the inclusion criteria and who volunteered to participate in the study, who applied to the Neurology outpatient clinic of the Medical Faculty Hospital will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of Respiratory Muscle Strength | baseline
  Maximum inspiratory (MIP) and expiratory pressures (MEP) are measurements of pressures against the closed airway to assess the strength of respiratory muscles. MIP and MEP pressures are noninvasive tests that show indirect respiratory muscle strength. Spirometry device (Carefusion /Micro RPM) will be used to assess MIP and MEP. The maximum inspiratory and expiratory valve (shutter) that closes the airway during the maximum oral pressure measured during the maximum breath.
Evaluation of Exercise Capacity | baseline
  Exerise capacity of participants will assess with TUG and 10MWT tests. Time up and go test (TUG) assesses mobility, balance, walking ability and risk of falling. The test is performed by the person getting up from a chair, walking 3 meters, turning around himself, walking back to the chair and sitting again.
  Ten meter walk test (10MWT): In the test, the person is asked to walk at his / her normal speed within a pre-measured area of 10 meters. Two measurements are taken and the best value is recorded in meters per second (m / sec).
Evaluation of Fatigue | baseline
  Fatigue impact scale (FIS) and Fatigue severity scale (FSS) will be used. Fatigue impact scale (FIS) consists of forty questions. The first 10 items assess cognitive status, the second 10 items evaluate physical status, and the third 20 items evaluate psychological status. Each question is scored between 0 (no problem) and 4 (maximum problem). The highest score is 160. Higher scores show more fatigue.
  Fatigue severity scale (FSS) consists of 9 questions. Each question is evaluated with a scale of 1 to 7 points. 1 = Strongly disagree, 7 = Strongly agree. Minimum score 9, maximum score 63.High scores indicate fatigue.
Evaluation of Physical Activity Level | baseline
  International Physical Activiy Questionnaire (IPAQ) will be used. The long form of the IPAQ questionnaire is used to gather information about recreational activities such as home and field activities, occupational transport, sedentary activities. The calculation of the total score for the IPAQ long form includes the sum of time (minutes) and frequency (days) for all types of activity in all areas. Scoring is done according to activity (walking, moderate activity, severe activity). From these calculations, a score in MET-minutes is obtained. A MET-minute is calculated by multiplying the minute of activity performed by the MET score. MET-min x (person's body weight kg / 60 kg). The following values are used for the analysis of IPAQ data.
  - Walking = 3.3 MET - Moderate physical activity = 4.0 MET - Severe physical activity = 8.0 MET

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No